CLINICAL TRIAL: NCT06361667
Title: "Culture and Well-being: Art as Prescription Therapy ("Art on Prescription"), Promoting Social Cohesion and Harnessing the "Silver Economy"
Brief Title: Culture and Well-being: Art as Prescription Therapy ("Art on Prescription")
Acronym: AoP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KAVADIA ELENI (Other)
Responsible Party: Sponsor-Investigator, KAVADIA ELENI, Executive Secretariat, University Mental Health Research Institute, Athens, Greece
Organization: University Mental Health Research Institute, Athens, Greece (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/02.02.2024
Record Dates: First submitted 2024-03-26; First posted 2024-04-12 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Mental Health Issue; Anxiety Disorders; Depressive Disorder; Emotional Disorder; Schizophrenia; Autism
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Schizophrenia; Autistic Disorder | interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Intervention Model Description: We will follow standard practice for RCTs and apply an ANCOVA model to estimate the effects of treatment. The formalism is:
  y ~ b0 + b1xtreatment_group + b2xtime + b3xtreatment_groupxtime + covariates (1)
  Where, y is each outcome, b1-b3 are the regression coefficients and covariates denotes covariates at randomisation (DETERMINE)
  The inference of interest for the model concerns b3, the interaction term, as we posit that there will be a difference in slopes between the treatment groups.
  The inference is going to happen via an estimation of the t-statistic, defined as follows"
  t = b3/SE (2)
  Where SE is the standard error for coefficient b3
  t > 1.96 (3)
  And 1.96 is the critical value for statistical significance at alpha = 0.05.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (AG) (Experimental): This arm will receive the arts intervention (any of the arts interventions).
  Interventions: Other: Arts
- Waitlist Control (WL) (Placebo Comparator): This arm will be the waitlist control and after 3 months it will be active.
  Interventions: Other: Arts

INTERVENTIONS:
Other: Arts — Arts (music, cinema, dance).
  Other Names: Art as Prescription Therapy

SUMMARY:
Stratified randomised controlled trial with two arms: arts intervention (any of the arts interventions, see list), which we call here Active Group (AG) vs waitlist control (WL).

DETAILED DESCRIPTION:
Design:

Stratified randomised controlled trial with two arms: arts intervention (any of the arts interventions, see list), which we call here Active Group (AG) vs waitlist control (WL). Stratifying will happen at each site.

Invastigators want to measure AG and WL, then WL becomes AG after 3 months and both the initial AG and the WL. AG will be measured in exactly the same way for another 3 months.

AG for 3 months. Then goes into 3 month follow up. WL for 3 months. Then this group receives intervention and becomes AG and has measurements for 3 months as the AG did.

There will be a 2-month break between T3 and T4 due to summer vacation.

In the beginning, an open invitation to institutions of culture and mental health had been sent. Culture institutions i.e. Opera House, Contemporary Art Museum, National Theater etc. presented their action plans for interventional courses. Investigators did the connection between mental health and culture institutions.

Potential participants declared their preference for the interventional course such as dance, cinema etc. and they listed while an external investigator did the blind randomization into AG or WL group.

Frequency of Measurement:

The primary outcome will be measured at time points (for adults):

* T0: (before the randomisation; patient's personal data and demographics)
* T1: (before the start of the intervention for the active group or the entry into the study for the WL group)
* T2: 6 weeks (after the start of the intervention for the active group or the entry into the study for the WL group)
* T3: 12 weeks (after the start of the intervention for the active group or the entry into the study for the WL group) The secondary outcomes will be measured at time points 0 (T4) and 12 weeks (T5) for both AG and WL.

The primary outcome will be measured at time points (for children/adolescents):

* T0: (before the randomisation; patient's personal data and demographics)
* T1: (before the start of the intervention for the active group or the entry into the study for the WL group)
* T3: 12 weeks (after the start of the intervention for the active group or the entry into the study for the WL group) The secondary outcomes will be measured at time points 0 (T4) and 12 weeks (T5) for both AG and WL.

ELIGIBILITY:
Inclusion Criteria:

* age range: 10-99 years
* be able to communicate effectively in order to provide answers to questionnaires that he/she will be asked to complete
* be able to commit to monitoring the action
* be able to participate in the activity alone (unaccompanied, without a carer),
* be able to answer the questionnaires
* to have legal capacity

Exclusion Criteria:

* active dependency,
* patients that are not consistent in following pharmaceutical drugs,
* patients from different Patient Association which is not "affiliated" with a Mental Health Professional Therapist.

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | 3 months
  The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS). This tool was developed in order to measure mental wellbeing in the general population by Tennant et al. (2007). It consists of 14 items responding using a 5-point Likert scale from 1 (never) to 5 (all the time). The overall score is calculated by summing the responses for every item without reversing none. The minimum overall score ranges from 14 to 70. Higher scores indicate increased mental wellbeing. The scale has been widely used nationally and internationally for monitoring, evaluating projects and programmes and investigating the determinants of mental wellbeing. An efficient internal consistency was proven using Cronbach's alpha score which was 0.89 for the student sample and 0.91 for the general population sample. Also, test-retest reliability at one week was high (0.83). The Greek validation showed acceptable internal consistency (Cronbach's alpha score 0.90).
The Patient Health Questionnaire-9 (PHQ-9) | 3 months
  The Patient Health Questionnaire-9 (PHQ-9) is a questionnaire which measures depression and grade severity of symptoms in general medical and mental health settings using nine DSM-5 criteria for major depression within the last two weeks. PHQ-9 constructed by Kroenke et al. (2001) and validated in Greek by Hyphantis et al. (2011) is using a four-point Likert-type scale. After summing all responses (0=not at all, 3=nearly every day), scores range from 0 to 27, with higher levels indicating increased symptom severity (0-4 no to minimal; 5-9 mild; 10-14 moderate; 15-19 moderately severe; 20-27 severe). The internal reliability of the PHQ-9 was excellent, with a Cronbach's α of 0.89 in the PHQ Primary Care Study (Kroenke et al., 2001) and 0.82 in Greek validation (Hyphantis et al., 2011).
Generalised Anxiety Disorder Assessment (GAD-7) | 3 months
  The Generalised Anxiety Disorder Assessment (GAD-7) is provided to screen symptom severity for the four most common anxiety disorders (generalized anxiety disorder, panic disorder, social phobia and posttraumatic stress disorder). GAD-7 constructed by Spitzer et al (2006) and validated in Greek by Vogazianos et al (2022). It consists of 7 items. The GAD-7 score is computed by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and summing together the scores for the seven questions (scores range from 0 to 21). Higher levels indicate increased anxiety. There are cut-offs for severity of anxiety as: (i) score 0-4: Minimal Anxiety; (ii) score 5-9: Mild Anxiety; (iii) score 10-14: Moderate Anxiety; (iv) score greater than 15: Severe Anxiety. The internal consistency of the GAD-7 was excellent (Cronbach α = 0.92) (Spitzer et al., 2006).

SECONDARY OUTCOMES:
UCLA 3-item Loneliness Scale | 3 months
  The Revised UCLA Loneliness Scale-20 (UCLA-20) is a questionnaire which measures level of psychological loneliness experienced by a person. UCLA-20 constructed by Russel et al. (1980) and validated in Greek by Anderson & Malikiosi-Loizos (1992). The internal reliability of the UCLA-20 was excellent, with a Cronbach's α of 0.94 (Russel et al., 1980) and 0.89 in Greek validation (Anderson & Malikiosi-Loizos, 1992). This long scale was shortened to 3 questions (UCLA 3-item Loneliness Scale) in order to be used in large surveys (Hughes et al., 2004). It is using a 3-point Likert-type scale (hard ever, some of the time, often). The scores can be added together to give a range of scores from 3 to 9. Higher scores mean most lonely (worse outcome).
The Strengths and Difficulties Questionnaire (SDQ) | 3 months
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioural screening tool for children and adolescents aged 2-17 years. PHQ-9 constructed by Goodman (2001) and validated in Greek by Gomez et al. (2021) is using a 3-point Likert-type scale ("not true," "somewhat true", "certainly true"). SDQ consists of 25 positive and negative items. These 25 items are divided between 5 scales: (i) emotional symptoms (5 items), (ii) conduct problems (5 items), (iii) hyperactivity/inattention (5 items), (iv) peer relationship problems (5 items), (v) prosocial behaviour (5 items). "Somewhat true" is always scored as 1 but the scoring of "not true" and "certainly true" varies and score 0 or 2. The total difficulties score is generated by summing the cores form all the scales except the prosocial scale. The final score can be ranged from 0 to 40. Higher scores mean most difficulties (worse outcome). Cronbach's alpha of the original study for all scales ranged from 0.35 to 0.64.

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Stefanis, PhD, Principal Investigator — University Mental Health Research Institute, Athens, Greece
Locations (1):
- Eleni Kavadia, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-03-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT06361667/Prot_001.pdf
  • Statistical Analysis Plan (2024-12-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT06361667/SAP_002.pdf